CLINICAL TRIAL: NCT04130867
Title: Defining Novel Pharyngeal Pressure Metrics to Predict Dysphagia Treatment Outcomes and Clinical Prognosis Using High-resolution Manometry
Brief Title: Rehabilitation Manometry Study
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-0576; A539770 (Other: UW Madison); SMPH/SURGERY/SURGERY*OT (Other: UW Madison); Protocol Ver 0.06, 1/16/2021 (Other: UW Madison)
Record Dates: First submitted 2019-10-15; First posted 2019-10-18 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Oropharyngeal Dysphagia
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group A: Swallow Therapy Oropharyngeal Strengthening: Participants receiving any standard of care swallow therapy with oropharyngeal strengthening as the primary goal
  Participants will undergo pHRM, videofluoroscopy (VF), diet assessment, functional reserve tests, and patient--reported outcome questionnaires at 3 standardized time points: baseline, 4 to 6 weeks (mid therapy), and 10 to -12 weeks (post -therapy)
  Interventions: Procedure: pHRM; Procedure: VFSS
- Group B: Surgical Treatment Esophageal Sphincter: Participants receiving surgical treatment for relief of upper esophageal sphincter outlet obstruction.
  Participants will undergo pHRM, videofluoroscopy (VF), diet assessment, functional reserve tests, and patient--reported outcome questionnaires at 3 standardized time points: baseline, 4 to 6 weeks (mid therapy), and 10 to -12 weeks (post therapy)
  Interventions: Procedure: pHRM; Procedure: VFSS
- Group C: Healthy Controls: Healthy controls (n=50) will also undergo data collection at parallel time points, without completion of a treatment paradigm.
  Interventions: Procedure: pHRM; Procedure: VFSS

INTERVENTIONS:
Procedure: pHRM — Pharyngeal high--resolution manometry (pHRM) provides direct and objective measurement of pressure changes in the pharynx that characterize basic mechanisms of swallowing.
Procedure: VFSS — Videofluoroscopic Swallow Study (VFSS) enables real-time visualization of bolus flow during swallow movement.

SUMMARY:
Oropharyngeal dysphagia, or difficulty swallowing, is a devastating condition that affects physiological and psychosocial functioning in 1 in 25 adults. Many dysphagia treatments exist, but our ability to adequately measure treatment outcomes is limited. Pharyngeal high-resolution manometry (pHRM) directly measures swallowing pressures, providing an objective measurement of physiology that characterizes the basic mechanisms of swallowing. pHRM is well-poised to measure outcomes of dysphagia treatments due to its direct, objective, and reproducible measures of swallowing function.

This proposed project will address a central hypotheses that objective swallowing measures (including (pHRM) will reveal treatment-mediated swallowing changes, will align with patient-reported outcome measures, and will be able to predict who will benefit from treatment. The investigators will follow a cohort of participants with oropharyngeal dysphagia as they undergo either pharyngeal strengthening therapy or relief of upper esophageal sphincter outlet obstruction at three time points: baseline, mid-treatment (4-6 weeks) and post-treatment (10-12 weeks). The investigators will compare participants to healthy controls using pHRM, videofluoroscopy, diet assessment, functional reserve tests, and patient-reported outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Pathological Group

  * Must have dysphagia as diagnosed by a licensed and certified otolaryngologist, gastroenterologist, or speech-language pathologist AND must have a dysphagia treatment plan that includes one of the following primary goals:

    * Therapy to strengthen oropharyngeal musculature
    * Medical or surgical management to relieve an obstruction at the upper esophageal sphincter
  * Must agree to comply with swallowing assessment, including interview and manometry
  * Must sign the Informed Consent form approved by the Health Sciences Institutional Review Board of the University of Wisconsin
* Normal Group

  * Having no swallowing disorders
  * Must agree to comply with swallowing assessment, including interview and manometry
  * Must sign the Informed Consent form approved by the Health Sciences Institutional Review Board of the University of Wisconsin.\

Exclusion Criteria:

* Pathological Group

  * Therapeutic management plan already initiated prior to recruitment
  * Therapy goals including only improvement of swallowing coordination
  * Developmental disability, dementia, cognitive dysfunction, or difficulty comprehending instructions
  * Positive history of allergic response to topical anesthetic
  * Allergy to food relevant to study participation (e.g. lactose intolerance)
* Normal Group

  * Known swallowing disorder
  * Developmental disability, dementia, cognitive dysfunction, or difficulty comprehending instructions
  * Positive history of allergic response to topical anesthetic
  * Allergy to food relevant to study participation (e.g. lactose intolerance)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 300 adults will be recruited to participate in the study. Participants will include 250 patients with heterogeneous causes of dysphagia undergoing active swallowing treatment and 50 age- and sex-match control participants with healthy swallow function. Participants will be stratified into the following goals of swallowing rehabilitation: Group A) Pharyngeal strengthening (n=125); and Group B) Relief of upper esophageal sphincter (UES) dysfunction or pharyngeal outlet obstruction (n=125). Classification will be based on clinician-driven diagnoses and treatment goals based on standard of care evaluation. The control group of healthy individuals will be Group C (n=50).
  Participants' age may range from 18-99 years old; as dysphagia is more frequent in the elderly, the sample will most likely include individuals age 60 and over.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2020-11-11 (Actual); Primary Completion 2021-04-21 (Actual); Study Completion 2021-04-21 (Actual)

PRIMARY OUTCOMES:
Change in pHRM from Baseline | up to 3 months
  pHRM data collected from the 250 adults undergoing dysphagia treatment and 50 healthy controls at three time points (baseline, mid-treatment, and post-treatment) will be used.
Change in Sydney Swallowing Questionnaire between timepoints | baseline, mid-treatment 4-6 weeks, post-treatment 10-12 weeks
  The Sydney Swallowing Questionnaire is a 17-item inventory scored on a visual analog scale (VAS) (with the exception of Q12) developed to measure symptomatic severity of pharyngeal dysphagia. Each VAS is 100 mm, where the left side of the scale is lesser symptoms and the right hand of the scale is increased symptoms. Scoring is measured in distance (mm) from the left. Maximum range in the scoring is 0 - 1700, the higher the score, the more severe the symptoms.
Change in Eat Assessment Tool Score between timepoints | baseline, mid-treatment 4-6 weeks, post-treatment 10-12 weeks
  The Eat Assessment Tool is a 10-item survey where each item is scored 0-4 where 0 is no problem and 4 is severe problem. The total range in score is 0-40 where higher scores indicate increased severity of symptoms.
Change in Hand Grip Strength Test between timepoints | baseline, mid-treatment 4-6 weeks, post-treatment 10-12 weeks
  Participants will squeeze a dynamometer at maximum pressure 3 times and hold for 5 seconds each. 10 seconds rest will be given between each trial.
Change in Maximum Isometric Pressure between timepoints | baseline, mid-treatment 4-6 weeks, post-treatment 10-12 weeks
  The Iowa Oral Pressure Instrument (IOPI) will be used to measure maximum isometric pressure. IOPI will be used to evaluate anterior and posterior maximal isometric tongue-pressures. A small (3.5 cm long and 4.5 cm in diameter) air-filled plastic pressure bulb will be placed in the mouth at two different positions: directly posterior to the incisors and at the posterior oral tongue. Participants will be asked to squeeze the bulb against the roof of the mouth with maximal effort and to perform saliva swallows. Three tasks in each position will be recorded and participants will rest for 10 seconds between each trial.
Change in Dietary Assessment between timepoints | baseline, mid-treatment 4-6 weeks, post-treatment 10-12 weeks
  Participants will undergo diet assessment by using International Dysphagia Diet Standardisation Initiative Framework. This framework defines and scores food textures/consistencies for participants with dysphagia. Liquids are scored 0-4 where 0 is thin and 4 is extremely thick. Foods are scored from 3-7 where 3 is liquidized food and 7 is regular food.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy McCulloch, MD, FACS, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No